CLINICAL TRIAL: NCT05345600
Title: A Pilot Randomized Trial Comparing the Use of MILTA vs Placebo for the Management of Pain Related to Perineal Scars Following Delivery
Brief Title: MILTA vs Placebo Use Comparison for the Management of Pain Related to Perineal Scars Following Delivery
Acronym: MILTADoIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2021_843_0049
Record Dates: First submitted 2022-03-22; First posted 2022-04-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Perineal Scars; Delivery Complication; Episiotomy; Pain; Treatment
Keywords: Perineal scars; Delivery Complication; episiotomy; Pain; treatment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MILTA (Experimental): The MILTA® uses photons which are emitted with low intensity in the visible and near infrared combining 5 physical principles to reduce pain
  Interventions: Other: MILTA probe
- placebo (Placebo Comparator)
  Interventions: Other: placebo probe

INTERVENTIONS:
Other: MILTA probe — Each woman will be included within the 6h after delivery (to ensure at least 2 days with the treatment / placebo). Once the written informed consent is obtained, the patient will be randomized in one of the 2 groups ("MILTA" or "Placebo"): 2 sessions are planned (the first one between 6h and 24h after delivery and the second one day after the first session). The woman will be lying on an exam bed. After a skin cleansing, the MILTA probe covered with a specific single use protection will be placed facing the scar. A 10-min session will include 5 min with the "analgesia mode" on followed with 5 min with the "healing mode" on in the MILTA group. For the placebo group, the procedure will be identical, with the probe switched OFF. To ensure that the red light is observable in the bedroom in both groups, a second probe will be used, facing the ceiling of the exam bedroom (and not the woman) for the 10 minutes of the procedure.
  Arms: MILTA
Other: placebo probe — Each woman will be included within the 6h after delivery (to ensure at least 2 days with the treatment / placebo). Once the written informed consent is obtained, the patient will be randomized in one of the 2 groups ("MILTA" or "Placebo"): 2 sessions are planned (the first one between 6h and 24h after delivery and the second one day after the first session). The woman will be lying on an exam bed. After a skin cleansing, the MILTA probe covered with a specific single use protection will be placed facing the scar. A 10-min session will include 5 min with the "analgesia mode" on followed with 5 min with the "healing mode" on in the MILTA group. For the placebo group, the procedure will be identical, with the probe switched OFF. To ensure that the red light is observable in the bedroom in both groups, a second probe will be used, facing the ceiling of the exam bedroom (and not the woman) for the 10 minutes of the procedure.
  Arms: placebo

SUMMARY:
The incidence of perineal scars after a pregnancy is high, either related to an episiotomy or to spontaneous perineal tears. These perineal scars can result in acute pain but also in chronic pain for some women. Medical treatment includes level 1 and 2 analgesics and, even for a few women, level 3 analgesic.

The MILTA® uses photons which are emitted with low intensity in the visible and near infrared combining 5 physical principles to reduce pain : 1- The NPCL (Nano-Pulsed Cold Laser) emissions in coherent infrared light, at 905 nanometers; 2- Non-coherent emissions, pulsed by trichromatic RGB CSM diodes (400 to 650 nm); 3- Continuous non-coherent infrared emission monochromatic diodes at 905 nm; 4- A constant circular magnetic field (200 millitesla) equivalent to the terrestrial magnetic field and 5- The effect of magnetic tunnel which potentiates the light propagation. MILTA® treatment has been shown to be effective in various managements of pain, but has never been used in pain related to perineal scars.

This randomized controlled trial aims at assessing MILTA vs placebo to reduce pain related to perineal scars after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* vaginal delivery less than 24h before inclusion
* perineal scar with pain assessed as > 3/10 with a numerical scale
* 18-years-old or older
* registration to the French medical system
* speaking and writing French
* written informed consent signed

Exclusion Criteria:

* woman under 18-years-old
* woman under law liberty restriction
* women unable to understand the written informed consent
* no written informed consent signed
* previous perineal surgery
* delivery with a caesarian section
* vaginal delivery with no perineal scar
* vaginal delivery with infected perineal scar
* women with restrictions for the use of level 1 analgesic
* women requiring level 2 or 3 analgesics for other reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 110 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2025-11-23 (Estimated)

PRIMARY OUTCOMES:
pain level | day 3
  Pain Level will be determined with EQ-5D instrument. The EQ-5D index scores were derived from the current UK tariff, which has a maximum value of 1 and a minimum value of -0.59.
  EQ-5D comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No